CLINICAL TRIAL: NCT06972030
Title: The Effect of Motivational Interviewing-Based Training on Peer Bullying, Social Exclusion and Aggression in Secondary School Students
Brief Title: Motivational Interviewing-Based Training
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Muş Alparslan University (Other)
Responsible Party: Principal Investigator, Kamile çiftci, Lecturer, Muş Alparslan University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: Peer Bullying
Record Dates: First submitted 2025-03-24; First posted 2025-05-14 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Social Exclusion; Aggression; Bullying of Child
Keywords: Peer bullying; Aggression; Social exclusion; Motivational interviewing
MeSH Terms: conditions — Social Isolation; Aggression | interventions — Motivational Interviewing

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental group (Experimental): After the pre-test, motivational interview-based training consisting of six sessions will be applied to the students in the experimental group, once a week. A pre-test, post-test (after 6 weeks) and a control test will be applied to both groups. At the end of the training, the training materials will be shared with the students.
  Interventions: Behavioral: Motivational interviewing
- Control group (No Intervention): The researcher will not apply any intervention to the control group other than the individual coping methods they apply in their daily lives. The training materials will be shared with the control group students at the end of the training.

INTERVENTIONS:
Behavioral: Motivational interviewing — After the pre-test, motivational interviewing-based training consisting of six sessions, once a week, will be applied to the students in the experimental group. A pre-test, post-test (after 6 weeks) and control test will be applied to both groups. At the end of the training, training materials will be shared with the students.
  Arms: Experimental group

SUMMARY:
The middle school period is the period when children begin to experience physical, emotional and social development and try to adapt to psychological changes. In this age group, which is seen as a transition period, the child's academic success and acceptance by peers and friends are also important. The problems experienced during this period can continue in adulthood and children are more likely to experience loneliness, sleep disorders, depression, anxiety, eating disorders, low self-esteem, suicidal thoughts, absenteeism and a decrease in academic success. For this reason, early detection of risky behaviors that threaten children's health and evaluation of health promotion practices are very important issues for child health nursing.

In recent years, peer bullying, aggression and social exclusion have increased and continue to increase in the middle school period, also called early adolescence. For this purpose, a study was needed to identify the situation in middle school students and reduce this negativity. In this respect, it is thought that the study will contribute to the literature. In addition, if the hypotheses of the study are confirmed, it is expected that similar training will be provided in other schools and contribute to the reduction of risky behaviors.

The aim of this study is to determine the effects of motivational interviewing-based education on peer bullying, social exclusion and aggression in secondary school students and to offer suggestions for situations where deficiencies are observed based on the findings obtained.

DETAILED DESCRIPTION:
The universe of the study consists of 1 secondary school selected by simple random method from 39 secondary schools located in the city center affiliated to the Muş Provincial Directorate of National Education. G Power 3.1.9.7 program was used to determine the sample size for the study. The program used the ''A priori: compute required sample'' analysis method. Accordingly, when the first type error amount (α = 0.05) was taken at an effect size of 0.365 (Seyhan Şahin & Ayaz-Alkaya, 2024), it was determined that the number of people to be included in the study to reach 99% power was 60 (30 intervention, 30 control).

Experimental and control groups will be determined by simple random method among the students who accept to participate in the research. Pre-test will be applied to the students in the control group, post-test will be applied 6 weeks after the pre-test and control test will be applied 3 months after the post-test. 6-week motivational interview based training will be given to the students in the experimental group after the pre-test. Post-test will be applied at the end of the training and control test will be applied 3 months after the post-test. In the study, first the control group and then the experimental group will be included in the study..

ELIGIBILITY:
Inclusion Criteria:

* Being 12-13 years old
* Being in one of the 6th and 7th grades of middle school
* Having a high score on the ''Peer Bullying Determination Scale''
* Being willing to participate in the research
* Not having a communication barrier
* The student and their parents having signed the informed consent form.

Exclusion Criteria:

* Having a low score on the ''Peer Bullying Determination Scale''
* The volunteer not wanting to continue during the research
* Encountering any communication barriers during the research
* Answering the data collection forms incompletely or incorrectly

Ages: 12 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-06-15 (Estimated)

PRIMARY OUTCOMES:
EFFECTS OF MOTIVATIONAL INTERVIEWING-BASED EDUCATION GIVEN TO SECONDARY SCHOOL STUDENTS ON PEER BULLYING, SOCIAL EXCLUSION AND AGGRESSION | First, a pre-test will be applied to students in both the experimental and control groups. A post-test will be applied to students in the control group after 6 weeks and a control test will be applied 3 months after the post-test. No intervention will be
  In the study, motivational interview-based training will be applied as a nursing intervention. After receiving institutional permission, a pre-test will be applied to students who agree to participate in the study to determine peer bullying. Students whose total scale score is above the average level will be randomly selected and included in the study will be determined. The study will begin after both groups have signed an informed consent form (both students and parents). In collecting research data, the "Introductory Information Form", "Peer Bullying Determination Scale", "Social Exclusion Scale for Children (SESC)", and "Aggression Scale" will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Kamile ÇİFTCİ, Study Director — Muş Alparslan University
Locations (1):
- Mus Alparslan University, Muş, Muş, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ding N, Zhang X. Bullying Victimization and Quality of Life among Chinese Adolescents: An Integrative Analysis of Internet Addiction and Social Withdrawal. Int J Environ Res Public Health. 2022 Dec 17;19(24):16973. doi: 10.3390/ijerph192416973. PMID 36554856